CLINICAL TRIAL: NCT00543296
Title: Re-implantation of a Fluocinolone Acetonide Implant for Non-infectious Uveitis Affecting the Posterior Segment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013641
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2014-06

CONDITIONS: Uveitis
Keywords: uveitis; Cystoid Macular Edema (CME); fluocinolone acetonide; non-infectious uveitis affecting the posterior segment
MeSH Terms: conditions — Uveitis; Macular Edema | interventions — Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.59 mg Fluocinolone Acetonide implant (Experimental): 0.59 mg Fluocinolone Acetonide implant
  Interventions: Drug: 0.59 mg Fluocinolone Acetonide implant

INTERVENTIONS:
Drug: 0.59 mg Fluocinolone Acetonide implant — 0.59 mg Fluocinolone Acetonide implant
  Other Names: Retisert

SUMMARY:
The purpose of this study is to collect data on patients with severe uveitis that have required re-implantation of the sustained-release fluocinolone drug delivery device due to depletion of study drug in their previous implanted device.

DETAILED DESCRIPTION:
Purpose: To collect medical information on a sustained release drug delivery system that delivers the corticosteroid, fluocinolone acetonide, directly into the vitreous cavity of the eye. This system has the potential to maintain therapeutic drug levels in the eye while reducing systemic exposure to the drug to negligible levels. RetisertTM is the trade name for the intravitreal fluocinolone acetonide implant.

Hypothesis: The RetisertTM will be a safe and effective method to manage patients with severe uveitis

ELIGIBILITY:
Inclusion Criteria:

* Non-infectious intermediate, posterior or panuveitis
* Previous placement of fluocinolone acetonide implant with initial uveitis quiescence and subsequent recurrence of inflammation once implant depleted of drug

Exclusion Criteria:

* Infectious uveitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Jaffe, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of these 21 subjects, 14 subjects had recurrence of inflammation and were re-implanted
Period: Overall Study
Arm/Group | 0.59 mg Fluocinolone Acetonide Implant
Started | 21
Completed | 14
Not Completed | 7
Not completed — Physician Decision | 7

BASELINE CHARACTERISTICS:
Population: Of 21 consented subjects only 14 completed the 9 months follow-up in whom fluocinolone acetonide implants were replaced or who needed a second implant.
Arm/Group | 0.59 mg Fluocinolone Acetonide Implant
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With Inflammation Recurrence
Description: Number of eyes with inflammation recurrence
Time Frame: 5 years
Measure: Number; unit: eye with inflammation
Units Other Than Participants: Number of eyes implanted
Arm/Group | 0.59 mg Fluocinolone Acetonide Implant
Number analyzed (Participants) | 14
Number analyzed (Number of eyes implanted) | 17
eye with inflammation | 1

2. Secondary Outcome: Percentage of Eyes With Improvement in Visual Acuity
Description: Visual acuity was improved by two or more lines from baseline.
Time Frame: baseline to 52 weeks
Population: There were 14 participants studied with a total of 17 eyes implanted. Of the 17 eyes each could require separate adjunctive therapy
Measure: Number; unit: percentage of eyes improved
Units Other Than Participants: Number of eyes implanted
Arm/Group | 0.59 mg Fluocinolone Acetonide Implant
Number analyzed (Participants) | 14
Number analyzed (Number of eyes implanted) | 17
percentage of eyes improved | 45

3. Secondary Outcome: Number of Participant's Eye Requiring Adjunctive Therapy
Description: Adjunctive Therapy needed to control inflammation in the implanted eye
Time Frame: 5 years
Population: as for outcome 2
Measure: Number; unit: participant's eyes
Units Other Than Participants: Number of eyes implanted
Arm/Group | 0.59 mg Fluocinolone Acetonide Implant
Number analyzed (Participants) | 14
Number analyzed (Number of eyes implanted) | 17
participant's eyes
  Topical corticosteroids | 12
  SubTenon triamcinolone acetonide injection | 7
  Prednisone | 1
  Intravitreal triamcinolone acetonide injection | 4

4. Secondary Outcome: Number of Eyes With Increased Intraocular Pressure
Time Frame: 52 weeks
Measure: Number; unit: eyes
Units Other Than Participants: Number of eyes implanted
Arm/Group | 0.59 mg Fluocinolone Acetonide Implant
Number analyzed (Participants) | 14
Number analyzed (Number of eyes implanted) | 17
eyes | 2

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | 0.59 mg Fluocinolone Acetonide Implant
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.59 mg Fluocinolone Acetonide Implant (N=14)
Endophthalmitis (Infections and infestations) | 1 (1) — Endophthalmitis is a known risk of ocular surgery
Retinial Detachment (Eye disorders) | 1 (1) — Retinal Detachment is a known risk of ocular surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes